CLINICAL TRIAL: NCT07368673
Title: Comparative Effectiveness of Ruxolitinib Monotherapy Versus Its Combination With Tacrolimus and Corticosteroids in the Management of Vitiligo: A Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tayyaba Iqbal, DR tAYYABA iQBAL, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTF-8
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Vitiligo
Keywords: vitiligo, ruxolitinib, tacrolimus, janus kinase inhibitors, repigmentation
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: participants will be randomized into three parallel treatment arms recieving either topical ruxilitinib monotherapy or ruxolitinib in combination with topical tacrolimus or topical corticosteroids
Masking Description: this is an open label study in which participants and investigators are aware of treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group a (Other): ruxolitinib monotherapy
  Interventions: Drug: ruxolitinib cream
- group b (Other): ruxolitinib with tacrolimus
  Interventions: Drug: ruxolitinib cream
- group c (Other): ruxolitinib with corticosteriods
  Interventions: Drug: ruxolitinib cream

INTERVENTIONS:
Drug: ruxolitinib cream — ruxolitinib cream applied topically twice daily to affected area for 24 weeks

SUMMARY:
this randomized controlled trial aims to compare the effectiveness and safety of ruxolitinib monotherapy versus its combination with topical tacrolimus or topical corticosteroids in patients with non-segmental vitiligo involving less than 10% body surface area. A total of 120 adult patients will be randomized into three treatment groups and followed for 24 weeks. Treatment response will be evaluated using validated scoring systems including the Vitiligo Area Severity Index (VASI), Vitiligo European Task Force (VETF) staging, and Physician Global Assessment. The findings may help optimize topical treatment strategies for vitiligo.

DETAILED DESCRIPTION:
Vitiligo is an acquired autoimmune skin disorder characterized by selective destruction of melanocytes, resulting in depigmented macules and patches affecting the skin, hair, and mucosa. The condition affects approximately 0.5-2% of the global population and can occur in both genders equally. Beyond its cutaneous manifestations, vitiligo has a profound psychosocial impact, often leading to reduced self-esteem and impaired quality of life.

The pathogenesis of vitiligo is multifactorial, involving genetic susceptibility, oxidative stress, immune dysregulation, and melanocyte apoptosis. Increased reactive oxygen species play a pivotal role in triggering melanocyte damage, particularly in genetically predisposed individuals. Conventional therapies, including topical corticosteroids, calcineurin inhibitors, and phototherapy, often yield variable results with frequent relapse.

Ruxolitinib, a topical Janus kinase (JAK) inhibitor, represents a novel targeted therapy that modulates the JAK-STAT signaling pathway involved in inflammatory cytokine signaling. It has demonstrated promising efficacy and an acceptable safety profile in non-segmental vitiligo. While ruxolitinib monotherapy is effective, the potential synergistic benefits of combining it with other topical immunomodulators such as tacrolimus or topical corticosteroids remain insufficiently studied.

This randomized controlled trial is designed to compare the clinical effectiveness of ruxolitinib monotherapy with its combination therapy using tacrolimus or topical corticosteroids. The study will be conducted in the outpatient dermatology department at Dow University of Health Sciences, Karachi, over a period of six months.

A total of 120 adult patients aged 18-65 years with non-segmental vitiligo involving less than 10% body surface area will be enrolled. Participants will be randomly assigned into three groups:

Group A: Topical ruxolitinib cream twice daily Group B: Tacrolimus 0.1% ointment in the morning plus ruxolitinib cream at night Group C: Topical fluticasone 0.05% cream in the morning plus ruxolitinib cream at night Clinical assessments will be performed at baseline and at weeks 4, 8, 16, and 24. Treatment efficacy will be evaluated using the Vitiligo Area Severity Index (VASI), Vitiligo European Task Force (VETF) staging, and Physician Global Assessment scores. Safety will be assessed by monitoring adverse effects throughout the study duration.

The results of this study are expected to provide evidence regarding the comparative effectiveness and safety of combination topical therapy versus ruxolitinib monotherapy, potentially guiding improved treatment strategies for patients with vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* adult aged 18 to 65 years male or female patients non-segmental vitiligo vitiligo involving less then 10% body surface area willingness to provide written informed consent

Exclusion Criteria:

* pregnant or lactating females known hypersentivity to ruxolitinib, tacrolimus or topical corticosteriods current use of systemic immunosuppressive therapy use of biologic therapy or phototherapy within the previous 12 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
change in VASI score | baseline to week 24
  the VASI will be used to assess the extent and degree of depigmentation. change in total VASI score from base line will be calculated to evaluate treatment efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tayyaba iqbal, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of health sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared due to ethical, institutional and confidentiality considerations